CLINICAL TRIAL: NCT03436082
Title: Post-Market Surveillance With a Novel mHealth Platform
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Johnson & Johnson (Industry); Food and Drug Administration (FDA) (U.S. Federal Agency); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2000021455
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Gastrectomy; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Data from a mHealth platform after bariatric surgery: Patients that have undergone sleeve gastrectomy or gastric bypass will pilot test the use of the patient-led, smartphone based, mhHealth platform HUGO.
  Interventions: Device: A mobile health platform
- Data from a mobile health platform after atrial fibrillation: Patients that have undergone a catheter-based atrial fibrillation ablation will pilot test the use of the patient-led, smartphone based, mobile health platform HUGO.
  Interventions: Device: A mobile health platform

INTERVENTIONS:
Device: A mobile health platform — Patients pilot testing the smartphone based, mobile health platform called HUGO. Patients will also be given syncable devices to use that will provide additional insights into their health and health outcomes.Patients will be queried about specific symptoms related to their procedure at enrollment, one week post-procedure, at 4 weeks and again at 8 weeks.

SUMMARY:
This is a study to pilot the feasibility of using a novel patient-led, smartphone-based mobile health platform (Hugo) for real-world surveillance of outcomes of patients after they undergo a bariatric surgical procedure (either sleeve gastrectomy or gastric bypass) and catheter-based atrial fibrillation ablation

DETAILED DESCRIPTION:
The plan is to pilot test a novel patient-led, smartphone-based mobile health platform (called Hugo) for real-world surveillance of outcomes in 60 total patients after medical device use. Research associates will be recruiting patients before they undergo a bariatric surgical procedure (either sleeve gastrectomy or gastric bypass) and catheter-based atrial fibrillation ablation. Patients will then be queried about specific symptoms related to their procedure. Patients will also be given syncable devices to use that will provide additional insights into their health and health outcomes. This pilot project will engage patients to report outcomes while also synchronizing data from their electronic health records and pharmacy accounts to ascertain the ability of emerging mobile health technologies to aid in post-marketing surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* English-speaking
* Planned for either a bariatric surgical procedure (either sleeve gastrectomy or gastric bypass) or catheter-based atrial fibrillation ablation
* Participant is willing and able to read and sign consent and participate in study
* Participant has an email account and a mobile device (smartphone or tablet) able to download the necessary applications
* Participant is willing to use the mobile health platform and syncable devices (e.g. Fitbit Charge 2)
* Attending bariatric surgeon or electrophysiologist (as appropriate) concurs that patient is a candidate for enrollment

Exclusion Criteria:

Healthy patients

Patients who refuse participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient's eligibility will first be determined by the implanting physician who will be performing the catheter-based atrial fibrillation ablation or bariatric surgical procedure (either sleeve gastrectomy or gastric bypass). The criterion used will simply be the cardiac electrophysiologist stating that the patient is being seen pre-procedurally for catheter ablation of atrial fibrillation or the bariatric surgeon stating that the patient is being seen pre-operatively for sleeve gastrectomy or gastric bypass.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ross, MD, Principal Investigator — Yale University; Sanket Dhruva, MD, Principal Investigator — Yale University; Nilay Shah, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dhruva SS, Ross JS, Akar JG, Caldwell B, Childers K, Chow W, Ciaccio L, Coplan P, Dong J, Dykhoff HJ, Johnston S, Kellogg T, Long C, Noseworthy PA, Roberts K, Saha A, Yoo A, Shah ND. Aggregating multiple real-world data sources using a patient-centered health-data-sharing platform. NPJ Digit Med. 2020 Apr 20;3:60. doi: 10.1038/s41746-020-0265-z. eCollection 2020. PMID 32352038
- [Derived] Bartlett VL, Ross JS, Shah ND, Ciaccio L, Akar JG, Noseworthy PA, Dhruva SS. Physical activity, patient-reported symptoms, and clinical events: Insights into postprocedural recovery from personal digital devices. Cardiovasc Digit Health J. 2021 Jul 3;2(4):212-221. doi: 10.1016/j.cvdhj.2021.06.002. eCollection 2021 Aug. PMID 35265911

RESULTS

PARTICIPANT FLOW:
Groups:
- Bariatric: (Sleeve Gastrectomy/Roux-en-Y)
- AF Ablation: Atrial Fibrillation Ablation
Period: Overall Study
Arm/Group | Bariatric | AF Ablation
Started | 30 | 30
Completed | 29 (Had procedure) | 30 (Had procedure)
Not Completed | 1 | 0
Not completed — Did not undergo procedure | 1 | 0

BASELINE CHARACTERISTICS:
Population: We enrolled a convenience sample of patients who were planning on undergoing either bariatric surgery (sleeve gastrectomy and gastric bypass) or catheter-based atrial fibrillation ablation at Yale-New Haven Hospital (YNHH) or the Mayo Clinic. 15 patients were enrolled for each procedure at each site, for a total of 60 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bariatric | AF Ablation | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 16 | 43
  >=65 years | 3 | 14 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (12.5) | 62.4 (10) | 55.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 7 | 18 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Disease-Specific PROMs Completed
Description: Disease-specific PROMs were collected using email notification to all patients over the course of the study. Disease-specific PROMs were emailed to patients at enrollment (preprocedure) and 1, 4, and 8 weeks post-procedure and were tailored to patients depending on the procedure they received. For each PROM, the date and time that it was emailed to patients, the time it was initiated, and the time at which the final response was received were all available.
Time Frame: 8 weeks
Population: Assessed for # disease-specific PROMs completed
Measure: Number; unit: # PROMs completed
Units Other Than Participants: # PROMs distributed
Arm/Group | Bariatric | AF Ablation
Number analyzed (Participants) | 29 | 30
Number analyzed (# PROMs distributed) | 75 | 73
# PROMs completed | 64 | 59
Statistical Analysis 1: Comparison: Bariatric vs AF Ablation; Test type: Other — We used Stata version 14.2 (StataCorp LP) to perform chi-square tests to compare syncing of the Fitbit device and response rate for the postprocedure recovery PROMs and disease-specific PROMs between patients in the bariatric surgery and atrial fibrillation ablation groups, using a p value < 0.05 to denote statistical significance; p = 0.04, Chi-squared

2. Primary Outcome: Number of Post-Procedure PROMs Completed
Description: Post-procedure PROMs were collected using email notification to all patients over the course of the study. Post-procedure PROMs were emailed to patients twice weekly for a total of 5 weeks post-procedure. Bariatric surgery patients were asked two questions: (1) if they had pain (yes/no) and, if yes, to rate their pain on a scale of 1-10 and (2) if they had an appetite (yes/no) and, if yes, to rate their appetite on a scale of 1-10. Atrial fibrillation ablation patients were asked about pain, as well as whether they had palpitations and, if yes, to rate both symptoms on a scale of 1-10. For each PROM, the date and time that it was emailed to patients, the time it was initiated, and the time at which the final response was received were all available.
Time Frame: 5 weeks
Population: Assessed for # PROMs completed
Measure: Number; unit: # PROMs completed
Units Other Than Participants: # PROMs distributed
Arm/Group | Bariatric | AF Ablation
Number analyzed (Participants) | 29 | 30
Number analyzed (# PROMs distributed) | 260 | 279
# PROMs completed | 203 | 237

3. Primary Outcome: Device Syncs
Description: Device syncs are operationally defined as the # of patients who synced their device at all required time points over the 8-week post-procedure period.
Time Frame: 8 weeks
Population: Assessed for # of device syncs
Measure: Number; unit: # patients who synced at all time points
Arm/Group | Bariatric | AF Ablation
Number analyzed (Participants) | 29 | 30
# patients who synced at all time points
  Fitbit | 17 | 14
  Disease-Specific (Withings Body Scale/Kardia Mobile) | 11 | 15
Statistical Analysis 1: Comparison: Bariatric vs AF Ablation; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.85, Chi-squared

4. Primary Outcome: Electronic Health Record Data Validation
Description: For EHR data, we validated the following components over 8 weeks follow-up: encounter date, encounter type, and encounter primary diagnosis. Specifically, we determined if encounters aggregated by the patient-centered health data sharing platform, Hugo, matched encounters listed in each patient's EHR.
Time Frame: 8 weeks
Population: Assessed for # times encounter date, encounter type, and encounter primary diagnosis matched between the data sharing platform, Hugo, and the patient's EHR
Measure: Number; unit: Number of matched records
Units Other Than Participants: Patient Records
Arm/Group | Bariatric | AF Ablation
Number analyzed (Participants) | 29 | 30
Number analyzed (Patient Records) | 106 | 115
Number of matched records
  Encounter Date | 105 | 110
  Encounter Type | 103 | 100
  Primary Diagnosis | 103 | 101

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Bariatric | AF Ablation
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

LIMITATIONS AND CAVEATS:
Enrolled a small number of patients (60) for a relatively short follow-up duration (8 weeks); EHR data for 5 patients were not observable in Hugo due to sync failure after portals were locked out from multiple incorrect password entries or an EHR upgrade; Stipends were provided to cover time and effort involved with study enrollment and participation and free personal digital devices, both of which may have enhanced engagement over the follow-up period; Did not examine quality of data obtained

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT03436082/Prot_000.pdf